CLINICAL TRIAL: NCT05625295
Title: Evaluation of the Implementation of Tele-dermatology, in Its Modality of Non-presential Inter-consultation, in the Province of Salamanca.
Brief Title: Tele-dermatology Non-presential (TeleDermaSA)
Acronym: TeleDermaSA
Status: Completed | Type: Observational
Sponsor: Fundacion para la Investigacion y Formacion en Ciencias de la Salud (Other)
Responsible Party: Principal Investigator, Luis Garcia Ortiz, PI, Fundacion para la Investigacion y Formacion en Ciencias de la Salud
Other Study IDs: 116
Record Dates: First submitted 2022-11-13; First posted 2022-11-22 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Teledermatology; Primary Care

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with non-face-to-face consultation: A sample of 500 patients who have undergone non-face-to-face consultation with dermatology
  Interventions: Other: data collection protocol in clinical history
- Patients with face-to-face consultation: A sample of 500 patients who have undergone face-to-face consultation with dermatology
  Interventions: Other: data collection protocol in clinical history

INTERVENTIONS:
Other: data collection protocol in clinical history — collection of data from the clinical history according to the established protocol

SUMMARY:
The purpose of the study is to evaluate the implementation of the Non-Face-to-Face Interconsultation of dermatology since it began to be used in August 2020 until August 2022 in the province of Salamanca (Spain)

DETAILED DESCRIPTION:
Design: cross-sectional descriptive study. Subjects: The unit of analysis will be the NPIs performed in dermatology since its implementation in August 2020 until the present time in the health area of Salamanca. To analyze the face-to-face consultations to analyze the differences. A random sample of 500 PNCIs and 500 face-to-face consultations will be extracted.

Measurements: To analyze the ICNP and face-to-face IC to dermatology registered in the computerized clinical history made in PC from Medora and registered in Jimena. To record the number of consultations, type of pathology referred, dermatology response time, discharges after assessment, face-to-face consultations required, delay time, treatment required, follow-up required or not, diagnostic coincidence, quality of the photographic image sent.

A differentiated analysis will be made according to the use or not of the dermatoscope, type of center (urban, semi-urban and rural), gender of the patients and age groups.

ELIGIBILITY:
Inclusion Criteria:

* The unit of analysis will be the PNCIs performed in dermatology from Primary Care, registered in Medora software, with its corresponding photographic file, and its response in Jimena software of the dermatology service, from June 2021 to June 2022, one year.

Exclusion Criteria:

-

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The unit of analysis will be the PNCIs performed in dermatology from Primary Care, registered in Medora software, with its corresponding photographic file, and its response in Jimena software of the dermatology service, from June 2021 to June 2022, one year. A random sample stratified by type of center (urban, semi-urban and rural) will be extracted.
  A control group of face-to-face consultations will be used, in a similar number (500) obtained randomly, and also stratified by type of center, which will be used to compare the information from the NCIs.
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Derivation rates per 10,000 h. | 1 year
  number of patients referred to the dermatology office

CONTACTS AND LOCATIONS:
Overall Officials: Luis G Garcia Ortiz, PhD, Study Director — FUNDACION INFOSALUD
Locations (1):
- Centro de Salud La Alamedilla, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sanchez-Martin E, Moreno-Sanchez I, Moran-Sanchez M, Perez-Martin M, Martin-Morales M, Garcia-Ortiz L. Store-and-forward teledermatology in a Spanish health area significantly increases access to dermatology expertise. BMC Prim Care. 2024 Jun 24;25(1):227. doi: 10.1186/s12875-024-02479-1. PMID 38914974